CLINICAL TRIAL: NCT06805136
Title: Tackling Youth Loneliness in Urban Areas: Measuring Feasibility, Acceptability, and Benefits of a Community-based Intervention.
Brief Title: Establishing Social Connections in Urban Areas: Evaluating a Community-based Programme
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QME24. 0657; APP19330 (Other: Economic and Social Research Council (ESRC) - UKRI)
Record Dates: First submitted 2025-01-09; First posted 2025-02-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Loneliness
Keywords: Loneliness; Young adults; Social interaction; Community intervention; Urban; Feasibility; Acceptability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based intervention group (Experimental): The participants in the community-based intervention group will be invited to attend weekly social activities over a period of 12 weeks. Participants must be committed to attend at least 8 activities during the 12 week period. Following the 12-week intervention period, the intervention group will enter a 6-week post-intervention period where they will no longer be encouraged to attend the activities to help understand the impact of stopping the intervention.
  Interventions: Behavioral: Community-based social interaction intervention
- Wait-list control (No Intervention): The participants allocated to the wait-list control will continue to receive any standard care they were receiving (e.g., National Health Services (NHS) services) during the 18-week trial. All participants will be eligible and able to access the community-based intervention as independent members once the trial ends (after 18 weeks).

INTERVENTIONS:
Behavioral: Community-based social interaction intervention — The intervention focuses on free or low-cost social interaction by offering community initiatives and activities, online spaces for interaction, and social events to young and working-age adults in London. Activities include but are not limited to social walks, bingo nights, board game afternoons and pub quizzes.
  Arms: Community-based intervention group

SUMMARY:
The aim of this study is to evaluate the feasibility and acceptability of a new community-based programme designed to tackle loneliness for young and working-age adults. The programme focuses on encouraging social interactions and connections through offering community initiatives and activities, online spaces for interaction, and free or low-cost social events for young adults. Further aims of this study are to determine the cost-effectiveness of the programme.

DETAILED DESCRIPTION:
Loneliness is associated with adverse mental and physical health outcomes. Most interventions are aimed at older adults even though young adults, including those of working-age, have been identified as being at-risk for persistent loneliness. This study aims to formatively evaluate the feasibility and acceptability of a community-based social interaction intervention. Therefore, the main objectives of this study are to:

1. Assess the feasibility and acceptability of the community-based intervention.
2. To determine the costs and effects related to the community-based intervention using quantitative feasibility study data and qualitative interviews with study participants.

In this mixed-methods two-arm randomised feasibility study with qualitative evaluation, participants will be randomly allocated to the community-based intervention over 12 weeks or to the wait-list control group. The intervention consists of weekly community social activities with the aim of reducing feelings of loneliness. Participants in the wait-list control group can continue any standard care or support they were receiving e.g. use of GP or mental health services. For both groups, online self-report assessments will take place at baseline (time 0, t0), 12-week follow-up (end of the intervention period; time 1, t1) and 6-weeks post intervention (18-weeks after baseline, time 2, t2). For the intervention group, an additional qualitative interview will be taken at the final timepoint (time 3, t3; 6 weeks post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40
* Reside in London
* Reports that they are some of the time or often lonely in response to a single questionnaire item ("How often do you feel lonely?)
* No prior interaction with the community-based intervention we are investigating
* Able to communicate in English sufficiently well to engage in qualitative interviews and complete the outcome measures and questionnaires.
* Available and willing to participate in the study for 18 weeks

Exclusion Criteria:

* Age < 20 or age >40.
* Resides outside of London.
* Does not report frequent levels of loneliness ("hardly ever or never" in response to single questionnaire item).
* Previously attended any event or is an existing member of the community-based programme that is forming the intervention arm.
* Unable to communicate even with communication support.
* Planned unavailability for >3 weeks during intervention and follow up periods.
* Participating in another research project related to loneliness.
* Reports current severe unstable health problems (mental or physical) or is deemed overburdened with respect to participating in research.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From enrollment to 6-weeks post-intervention (18 weeks total)
  To determine feasibility, we will record: (i) Number of participants that complete the screening stage. (ii) Number of eligible participants following the screening. (iii) Number of participants who consent to take part in the intervention. (iv) Number of participants randomised. (v) Number of participants who drop out and reasons offered for this. (vi) During the intervention: range and average number of sessions completed as a proportion of those offered. Data completeness for each questionnaire will be summarised at each time point.
Acceptability | 6-weeks post intervention
  Qualitative interviews will be conducted to explore participants' experiences of the intervention, barriers and facilitators, perceived active ingredients, potential benefits, and suggested changes. They will also seek to understand the reach, engagement, and benefits of the intervention by focusing on topics around engagement, tolerability, and safety. The interviews will be conducted with the intervention group and facilitated using topic guides.

SECONDARY OUTCOMES:
Loneliness | Start of the intervention (baseline), end of intervention follow-up (12-weeks), 6-weeks post intervention (18 weeks).
  The University of California Los Angeles (UCLA) loneliness scale. The UCLA loneliness scale consists of 20 questions related to loneliness, including how often you 'lack companionship', 'feel left out', or 'feel isolated from others'. Higher scores indicate greater levels of loneliness
Wellbeing | Start of the intervention (baseline), end of intervention follow-up (12-weeks), 6-weeks post intervention (18 weeks).
  The short version of the Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS). The SWEMWBS measures mental wellbeing using 7 statements with a recall period of 2 weeks. Higher scores indicate higher positive mental wellbeing.
Social connectedness | Start of the intervention (baseline), end of intervention follow-up (12-weeks), 6-weeks post intervention (18 weeks).
  The Social Connectedness Scale (SCS). This SCS scale measures connectedness using 20 items measuring belongingness, on a 6-point Likert scale.
Health Related Quality of Life | Start of the intervention (baseline), end of intervention follow-up (12-weeks), 6-weeks post intervention (18 weeks).
  The European Quality of Life 5 Dimensions 5 Level version (EQ-5D-5L) has five dimensions, each dimension has five levels of response. The dimensions cover mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores are used to obtain utility values where one is perfect health, 0 represents death, and negative scores reflect health states worse than death.
Capability | Start of the intervention (baseline), end of intervention follow-up (12-weeks), 6-weeks post intervention (18 weeks).
  ICEpop CAPability measure for Adults (ICECAP-A). This tool assesses five capabilities covering feeling settled/secure, love/friendship/support, being independent, achievement/progress, and enjoyment/pleasure. Each capability has four levels of response.
Client Service Receipt Inventory | Start of the intervention (baseline), end of intervention follow-up (12-weeks), 6-weeks post intervention (18 weeks).
  Client Service Receipt Inventory (CSRI) captures health and social care resource utilisation. These will be recorded over a 6-week period. Questions will include frequency of resource use in primary, community, and secondary care, medications, and employment status. Health and social care resource use will be used, combined unit costs, to evaluate the cost of healthcare resources used by each group (intervention and control) Unit costs will be obtained from the Unit Costs of Health and Social Care, supplemented with the National Reference Costs.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - In the community in London, England, London
  - Youth Resilience Unit, Wolfson Institute of Population Health, Queen Mary University of London, London

IPD SHARING:
Plan to Share IPD: Yes
Participants' anonymised data may be shared with other research scientists for the purposes of research and knowledge.
Supporting Information: Study Protocol
Time Frame: Fully anonymised and non-identifiable study data will be available 6 months following the project's end, and will be kept by the PI for at least 10 years in the approved long-term repository in the UK.
Access Criteria: Participants' anonymised data may be shared with other research scientists for the purposes of research and knowledge. This data will not be able to be traced back to participants. The datasets will be available upon request from Professor Jennifer Lau, who is the lead researcher.

REFERENCES:
- [Background] Al-Janabi H, Flynn TN, Coast J. Development of a self-report measure of capability wellbeing for adults: the ICECAP-A. Qual Life Res. 2012 Feb;21(1):167-76. doi: 10.1007/s11136-011-9927-2. Epub 2011 May 20. PMID 21598064
- [Background] Shah N, Cader M, Andrews B, McCabe R, Stewart-Brown SL. Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS): performance in a clinical sample in relation to PHQ-9 and GAD-7. Health Qual Life Outcomes. 2021 Nov 24;19(1):260. doi: 10.1186/s12955-021-01882-x. PMID 34819104
- [Background] Russell D, Peplau LA, Ferguson ML. Developing a measure of loneliness. J Pers Assess. 1978 Jun;42(3):290-4. doi: 10.1207/s15327752jpa4203_11. PMID 660402
- [Background] Bryan BT, Thompson KN, Goldman-Mellor S, Moffitt TE, Odgers CL, So SLS, Uddin Rahman M, Wertz J, Matthews T, Arseneault L. The socioeconomic consequences of loneliness: Evidence from a nationally representative longitudinal study of young adults. Soc Sci Med. 2024 Feb 22;345:116697. doi: 10.1016/j.socscimed.2024.116697. Online ahead of print. PMID 38490911
- [Background] Eager S, Johnson S, Pitman A, Uribe M, Qualter P, Pearce E. Young people's views on the acceptability and feasibility of loneliness interventions for their age group. BMC Psychiatry. 2024 Apr 23;24(1):308. doi: 10.1186/s12888-024-05751-x. PMID 38654301